CLINICAL TRIAL: NCT05459090
Title: Functional Study of Inhibitory and Excitatory Neurotransmission in the Nervous Tissue Resected From Human Brain: Understanding New Molecular Mechanisms and Discovering New Therapeutic Targets to Cure Drug-resistant Epilepsy.
Brief Title: Functional Study of Inhibitory Neurotransmission in the Human Epileptic Brain.
Status: Recruiting | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Katiuscia Martinello, Researcher, PhD, Neuromed IRCCS
Other Study IDs: LES-001
Record Dates: First submitted 2022-07-12; First posted 2022-07-14 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Drug Resistant Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with drug resistant epilepsy: All patients with drug-resistant epilepsy who undergo neurosurgical resection of the epileptic focus.
  Interventions: Other: ex-vivo study

INTERVENTIONS:
Other: ex-vivo study — ex-vivo experiments in tissue slices obtained from biopsies
  Other Names: ex-vivo neuron-neuron communication

SUMMARY:
Epilepsy is a neurological condition that afflicts 1% of the world population. 30% of patients become drug-resistant to classic antiepileptic treatment and only a small percentage, 5%, can undergo a neurosurgical resection of epileptic focus and recover almost completely from symptoms. To date, an imbalance between inhibitory and excitatory neurotransmission has been well accepted as the main root cause of epilepsy. A better understanding of the molecular mechanisms of this can lead to developing new therapeutic strategies. The investigators of the project want to describe the functional alteration of GABA- A receptor, the main actor of inhibitory neurotransmission in the central nervous system and characterize its subunit composition in the epileptic foci of patients with temporal lobe epilepsy. The authors, also, want to modulate, by means of selective neuroactive molecules, the function of this receptor to increase the inhibitory tone in the epileptic brain.

DETAILED DESCRIPTION:
The project presents 3 aims:

1. Characterization of macroscopic GABA-A mediated currents evoked by the specific agonist, muscimol, in presence of selective negative and positive allosteric modulators to identify the subunit composition.
2. Functional characterization of synaptic GABA-A mediated currents recorded from hippocampal and cortical pyramidal neurons by using pharmacological tools.
3. After the acquired knowledge of aims 1) and 2), promotion of the increase of inhibitory tone in epileptic tissue, enhancing the GABA release from interneurons onto principal cells, by stimulation of other neurotransmitter systems present in the brain: cholinergic system, serotonergic system, and dopaminergic system.

Experimental design:

AIM1 WP1.1: Patch-clamp recordings of whole-cell GABA-A mediated currents from pyramidal and interneurons evoked by muscimol, perfusing the slices with positive allosteric modulators such as diazepam or nitrazepam, that are selective for apha1/alpha2 subunits GABA-A containing receptors or phenobarbital selective for alpha4/alpha6 subunits GABA-A containing receptors.

WP 1.2: Patch-clamp recordings of whole-cell GABA-A mediated currents from pyramidal and interneurons evoked by muscimol, perfusing the slices with negative allosteric modulators such as BetaCCT, which is selective for apha1/alpha2 subunits GABA-A containing receptors or L655,708 and Furosemide that are selective for alpha4/alpha6 subunits GABA-A containing receptors.

AIM2 WP2.1: Patch-clamp recordings of spontaneous and evoked GABA-A synaptic currents from interneurons and pyramidal cells and their modulation by the same pharmacological tools as in Aim 1, WP2.2: Patch-clamp recordings of spontaneous and evoked glutamatergic synaptic currents from interneurons and pyramidal cells and their modulation by the GABA positive and negative allosteric modulators.

AIM3 WP 3.1:Increase of GABA release, by recording spontaneous currents in pyramidal neurons, modulating, by means of allosteric modulators the cholinergic, dopaminergic, and serotonergic receptors.

Methodologies and statistical analyses:

During the neurosurgical approach, 1 cube cm of total biopsic tissue will be used for ex-vivo experiments.Transversal neocortical or hippocampal slices (350 μm thickness ) will cut in glycerol-based artificial cerebrospinal fluid (ACSF) with a vibratome (Leica VT 1000S) immediately after surgical resection. Slices will be placed in a slice incubation chamber at room temperature with oxygenated ACSF and transferred to a recording chamber within 1-24 h after slice preparation. Whole-cell patch-clamp recordings will be performed on pyramidal cells or interneurons at 22-25°C.

Both excitatory and inhibitory spontaneous or miniature post synaptic currents will be recorded using a Multiclamp 700B amplifier (Axon Instruments, Foster City, CA, USA), -70 mV holding potential, in the presence of TTX, 1 microM, CNQX, 20microM and (AP5, 40microM to block sodium currents, AMPA, kainate and NMDA receptors respectively or in presence of bicuculline (20 microM) and CGP55845 (50nM) to block GABA -A and -B receptors when necessary. Patch pipettes will be filled with the intracellular solution containing: 140 mM KCl, 10 mM HEPES, 0.5 mM EGTA and 2 mM Mg-ATP (pH 7.35, with KOH). Input and series resistances will be monitored during the experiments every five minutes, and >10% changes excluded the cell from further analysis. GABA-A receptor agonist or antagonist will be administrated to the cells by perfusion in the bath solution for 10 minutes.

Chemicals and Solutions. ACSF will have the following composition: 125 mM NaCl, 2.5 mM KCl, 2 mM CaCl2, 1.25 mM NaH2PO4, 1 mM MgCl2, 26 mM NaHCO3, 10 mM glucose, 0.1 mM Na-pyruvate (pH 7.35). Glycerol-based ACSF solution will contain 250 mM glycerol, 2.5 mM KCl, 2.4 mM CaCl2, 1.2 mM MgCl2, 1.2 mM NaH2PO4, 26 mM NaHCO3, 11 mM glucose, and 0.1 mM Na-pyruvate (pH 7.35).

Data analysis and statistics. The analysis of electrophysiological parameters will be performed with Clampfit 10 software (Axon Instruments, Foster City, CA, USA) by using a detection algorithm based on a sliding template. To characterize the currents it will be used: i) the rise time (estimated as the time needed for 10-90% increase of the peak current response); ii) the decay time (as the time needed for 90-10% decrease of peak current); iii) the mean charge of a single synaptic event, Q (measured as the time integral of the currents); vi) amplitude and v) frequency of synaptic events. Statistical comparisons between groups were made with the One Way ANOVA test (Shapiro-Wilk normality test; equal variance test) and all pairwise multiple comparisons with the Holm-Sidak method. The power of all performed tests was > 0.8 (alpha=0.05). P<0.05 was taken as significant. In case of failure of normality test or equal variance test, Kruskal-Wallis One Way ANOVA on ranks was used, with Dunn's method for pairwise comparisons.

To calculate the number of participants (n patients=n of cells) we use "The iterative method of Camussi et al., 1995." following the relation where n is the number of human neurons: n>2sigma^2 (z* alpha/D)^2, where sigma must be substituted with an estimate of sampling variance (s^2), alpha=0.05, z*alpha=-2, and D is the difference between treatments. With this consideration, 12 patients for each WPI previously described will be necessary. In total 60 patients will be involved in the study in 5 years.

.

ELIGIBILITY:
Inclusion Criteria:

Patients with drug-resistant temporal lobe epilepsy.

Exclusion Criteria:

* Patients suffering from Temporal lobe epilepsy caused by stroke, ischemia, cavernous angiomas, or meningiomas growth.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with drug-resistant TLE who undergo neurosurgery for resection of epileptic focus
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Composition of GABA-A receptors that modulate macroscopic currents | 24 months
  WP1.1- Slices of tissue obtained from 12 patients Tratment :diazepam or nitrazepam and phenobarbital
  WP 1.2:- Slices of tissue obtained from 12 patients Treatment: BetaCCT and L655,708 or Furosemide .
Modulation of synaptic transmission by GABA-A receptors PAMs and NAMs | 24
  WP2.1 Slices of tissue obtained from 12 patients
  Treatment: diazepam, phenobarbital, BetcCCt, and Furosemide, effect on inhibitory synaptic transmission
  WP2.2: Slices of tissue obtained from 12 patients Treatment: diazepam, phenobarbital, BetcCCt, and Furosemide, effect on excitatory synaptic transmission
Modulation of inhibitory synaptic transmission by cholinergic, dopaminergic and serotonergic PAMs. | 12
  WP 3.1 Slices of tissue obtained from 12 patients
  Based on results obtained in Primary Outcome 1 and 2 Treatment: PNU dFBr, mCPGB, or L-dopa, effect on inhibitory neurotransmission.

CONTACTS AND LOCATIONS:
Overall Officials: katiuscia Martinello, Biology, Principal Investigator — Neuromed IRCCS
Locations (1):
- IRCCS INM Neuromed, Pozzilli, Isernia, Italy

IPD SHARING:
Plan to Share IPD: No